CLINICAL TRIAL: NCT03421717
Title: The Effect of Peri-implant Surgery and Chair-side Supportive Post Surgical Peri-implant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Odd Carsten Koldsland, Associate professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Peri-implantitis
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Periimplantitis; Peri-implant Mucositis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: 6 month after surgical intervention, the population is randomly assigned to two parallel groups, receiving one of two maintenance programs - use of titanium curettes or chitosan brushes. Randomization was performed by pulling notes test/control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Maintenance treatment (test/control) was performed after the investigator left the room. Investigator did not have access to the registration forms where information regarding assignment (test/control) was noted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Treatment/maintenance of implants postsurgically performed by the use of chitosan brushes
  Interventions: Device: Chitosan brush
- Control (Active Comparator): Treatment/maintenance of implants postsurgically performed by the use of titanium curettes
  Interventions: Device: Chitosan brush

INTERVENTIONS:
Device: Chitosan brush — If inflammation (Bleeding on probing) and deep pockets (4 mm or more) is present at the control - maintenance is performed according to allocation
  Other Names: Titanium curettes

SUMMARY:
Peri-implantitis is defined as inflammation in the mucosa surrounding an oral implant with loss of supporting bone. The goals of peri-implantitis treatment are to resolve inflammation and to arrest the progression of disease. It is important to systematically gather information on the effect of surgical peri-implant treatment and to assess different protocols regarding chair-side maintenance of peri-implant tissue after surgery

The aims of this clinical investigation are to evaluate the clinical, microbiological and radiographic outcomes of surgical treatment of peri-implantitis and to evaluate the efficacy of 2 supportive treatment protocols based on the use of titanium cyrettes or by the use of a flexible, biodegradable chitosan brush. Furthermore, to evaluate the impact of this therapy on selected biochemical markers associated with chronic inflammation and bone tissue destruction.

DETAILED DESCRIPTION:
Little is known about the effect of chair-side maintenance of dental implants after peri-implantitits surgery. Traditionally, the maintenance has been performed by titanium curettes to remove microbiological deposits from the submucosal area.

The Labrida biodegradable brush is a novel debridement device intended for use on dental implants. The concept of using a biodegradable material is related to the suggested problems with leaving remnants on the treated implant surface which would be negative from a bone regenerative aspect. The use of a flexible brush relates to the access problems when treating dental implants both related to the threads as well as due to the prosthetic supra construction hindering access for debridement with regular instruments developed for teeth. The material used in the brush will be Chitosan which is a natural polysaccharide, chitosan (poly-N-acetyl glucosaminoglycan), which is a nontoxic and bioabsorbable (REK-approval 2012/791 polymer).

H0: It is possible to maintain peri-implant health after surgical peri-implantitis treatment. There is no short- or long term clinical or radiographical differences between patients surgically treated for peri-implantitis maintained by the use of titanium cyrettes or with the Labrida brush in chair-side supportive care

ELIGIBILITY:
Inclusion Criteria:

Overt peri-implantitis presenting at least one implant with;

* radiographic bone loss ≥ 2.0 mm
* bleeding on probing (BoP)

Main exclusion criteria:

* radiotherapy
* chemotherapy
* systemic long-term corticosteroid treatment
* pregnancy or nursing
* anatomical abnormalities
* history of previous treatment of peri-implantitis within 6 months after the screening
* American Society of Anesthesiologists (ASA) classification for assessing the fitness of patients before surgery > 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Inflammation control | 3 months
  Absence/presence of bleeding on probing and deep peri-implant pockets

SECONDARY OUTCOMES:
Progressive bone loss | 3 months
  Loss of attachment at the implant identified on radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Odd Carsten Koldsland, Ph.D, Principal Investigator — Institute of Clinical Odontology, Faculty of Dentistry, University of Oslo

IPD SHARING:
Plan to Share IPD: No
Data will be handeled by the investigators treating the patients and collecting data